CLINICAL TRIAL: NCT00269880
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled Trial Evaluating Clinical Outcomes Following Percutaneous Coronary Intervention in Patients Treated With an Abciximab Bolus Plus 12-Hour Infusion Given With Either Standard-Dose Weight-Adjusted Heparin or Low-Dose Weight-Adjusted Heparin
Brief Title: A Study Comparing the Efficacy and Safety of Abciximab, an Anti-Platelet Therapy, in Combination With Two Different Heparin Regimens in Patients Undergoing Percutaneous Coronary Intervention.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR006262
Record Dates: First submitted 2005-12-22; First posted 2005-12-26 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Angioplasty, Transluminal, Percutaneous Coronary
Keywords: Angioplasty, Transluminal, Percutaneous coronary
MeSH Terms: interventions — Heparin; Abciximab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Placebo and Standard Dose of Heparin (Placebo Comparator): Participants will receive bolus placebo followed by 12-hour infusion of placebo and bolus heparin at a dose of 100 units per kilogram of body weight.
  Interventions: Drug: Placebo; Drug: Heparin
- Abciximab and Low Dose of Heparin (Active Comparator): Participants will receive bolus abciximab at a dose of 0.25 milligram per kilogram (mg/kg) of body weight followed by 12-hour infusion of 0.125 microgram per kilogram per minute (mcg/kg/min) and bolus heparin at a dose of 70 units per kilogram of body weight.
  Interventions: Drug: Heparin; Drug: Abciximab
- Abciximab and Standard Dose Heparin (Active Comparator): Participants will receive bolus abciximab at a dose of 0.25 mg/kg of body weight followed by 12-hour infusion of 0.125 mcg/kg/min and bolus heparin at a dose of 100 units per kilogram of body weight.
  Interventions: Drug: Heparin; Drug: Abciximab

INTERVENTIONS:
Drug: Placebo — Placebo is administered as bolus or 12 hour infusion prior to index percutaneous coronary intervention.
  Arms: Placebo and Standard Dose of Heparin
Drug: Heparin — Heparin is administered as either high dose (100 units/kg of body weight) or low dose (70 units/kg of body weight) boluses.
Drug: Abciximab — Abciximab is administered as bolus followed by 12 hour infusion prior to index percutaneous coronary intervention.
  Arms: Abciximab and Low Dose of Heparin; Abciximab and Standard Dose Heparin

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of abciximab, an anti-platelet therapy, versus placebo in patients undergoing percutaneous coronary intervention when administered in combination with two different heparin regimens. Please see attached results.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled trial comparing the efficacy and safety of abciximab, an anti-platelet therapy, in combination with two different heparin regimens in patients undergoing percutaneous coronary intervention. Patients will be randomly assigned to one of three treatment groups: abciximab/low-dose weight-adjusted heparin, abciximab/standard-dose weight-adjusted heparin, or placebo/standard-dose weight-adjusted heparin. The primary outcomes of the study include the number of deaths, myocardial infarctions, or repeat revascularizations within 6 months, and the number of deaths, myocardial infarctions, or severe myocardial ischemia leading to urgent repeat percutaneous coronary intervention or urgent coronary artery bypass surgery within 30 days. Please see attached results.

Abciximab bolus plus 12-hour infusion with standard-dose weight-adjusted heparin; Abciximab bolus plus 12-hour infusion with low-dose weight-adjusted heparin; Placebo bolus plus 12-hour infusion with standard-dose weight-adjusted heparin

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for elective or urgent percutaneous coronary intervention with an FDA-approved device
* Having a target artery (native or graft) stenosis of 60% by visual estimation

Exclusion Criteria:

* Patients with unstable angina/non-Q-wave myocardial infarction meeting EPIC criteria within the previous 24 hours, or with acute Q-wave myocardial infarction meeting EPIC criteria with onset of chest pain within previous 24 hours
* With active internal bleeding, having a condition that may increase the risk of bleeding, or currently receiving administration of oral anticoagulants at the time of study entry
* With confirmed hypertension with systolic blood pressure >180 mm Hg or diastolic blood pressure >100 mm Hg
* Having had a percutaneous coronary intervention within the previous 3 months
* Having an unprotected left main coronary artery stenosis > 50%

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2792 (Actual)
Dates: Start 1995-02; Primary Completion 1995-12 (Actual); Study Completion 1995-12 (Actual)

PRIMARY OUTCOMES:
Death, myocardial infarction, or repeat revascularization within 6 months | up to 6 months
Death, myocardial infarction, or severe myocardial ischemia leading to urgent repeat percutaneous coronary intervention or urgent coronary artery bypass surgery within 30 days | Up to 30 Days

SECONDARY OUTCOMES:
Angiographic outcome; death, MI or target vessel revascularization within 6 months; death or MI within 6 months; health economic analyses | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.

REFERENCES:
- [Result] Lincoff AM, Mark DB, Tcheng JE, Califf RM, Bala MV, Anderson KM, Davidson-Ray L, Knight JD, Cabot CF, Topol EJ. Economic assessment of platelet glycoprotein IIb/IIIa receptor blockade with abciximab and low-dose heparin during percutaneous coronary revascularization: results from the EPILOG randomized trial. Evaluation in PTCA to Improve Long-term Outcome with abciximab GP IIb/IIIa blockade. Circulation. 2000 Dec 12;102(24):2923-9. doi: 10.1161/01.cir.102.24.2923. PMID 11113041
- [Result] Lincoff AM, Tcheng JE, Califf RM, Kereiakes DJ, Kelly TA, Timmis GC, Kleiman NS, Booth JE, Balog C, Cabot CF, Anderson KM, Weisman HF, Topol EJ. Sustained suppression of ischemic complications of coronary intervention by platelet GP IIb/IIIa blockade with abciximab: one-year outcome in the EPILOG trial. Evaluation in PTCA to Improve Long-term Outcome with abciximab GP IIb/IIIa blockade. Circulation. 1999 Apr 20;99(15):1951-8. doi: 10.1161/01.cir.99.15.1951. PMID 10208997
- [Result] EPILOG Investigators. Platelet glycoprotein IIb/IIIa receptor blockade and low-dose heparin during percutaneous coronary revascularization. N Engl J Med. 1997 Jun 12;336(24):1689-96. doi: 10.1056/NEJM199706123362401. PMID 9182212
- See also: A Study of Siltuximab (Anti-IL-6 Monoclonal Antibody) Effects on the QT Interval in Subjects with Monoclonal Gammopathy of Undetermined Significance, Smoldering Multiple Myeloma, or Indolent Multiple Myeloma — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=213&filename=CR017452_CSR.pdf